CLINICAL TRIAL: NCT05490888
Title: A Phase 1 Open Label Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PHIN-214 in Adults With Child Pugh A and B Cirrhosis
Brief Title: Single and Multiple Dose Escalation of PHIN-214 in Child-Pugh A and B Liver Cirrhotics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaIN (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHIN-001
Record Dates: First submitted 2022-07-28; First posted 2022-08-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis, Liver; Liver Fibrosis; Ascites Hepatic
Keywords: Terlipressin; Cirrhosis; Vasoconstrictor; Refractory Ascites
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- single dose of PHIN-214 (Experimental): Participants in Part 1 will receive one dose of PHIN-214 administered subcutaneously. Dose level will be assigned in ascending doses to observe initial safety and tolerability. A Safety Committee will review information from each patient and determine the dose level for the subsequent participants.
  Interventions: Drug: PHIN-214 Subcutaneous injection
- multiple daily dosing of PHIN-214 (Experimental): Participants in Part 2 will be trained to give themselves a daily dose of PHIN-214 at home by subcutaneous injection for 28-days. The dose level assigned to each participant will be determined by a Safety Committee after reviewing information from the last participants' experience and compilation of experiences on all previous participants. Dose level advancement will be guided throughout the study by the experiences and information collected from each participant.
  Interventions: Drug: PHIN-214 Subcutaneous injection

INTERVENTIONS:
Drug: PHIN-214 Subcutaneous injection — subcutaneous injection(s) with PHIN-214 terlipressin derivative
  Other Names: Terlipressin derivative

SUMMARY:
This 2-part study will evaluate PHIN-214 given as a single one-time dose (Part 1) and in multiple doses (given as daily doses for 28-days) (in Part 2). Specifically, this study evaluates PHIN-214, to determine the safety, tolerability, and pharmacokinetic effects of PHIN-214, and to establish the maximum tolerated dose or optimal beneficial dose in patients with Child Pugh A and B Cirrhosis.

DETAILED DESCRIPTION:
PHIN-214 action has similar actions as another medication called "terlipressin or TERLIVAZ®." Terlipressin has been shown to reduce portal hypertension, improve renal function, and induce natriuresis in cirrhotic patients with ascites without hepatorenal syndrome (HRS). It is approved in several countries including the US for the treatment of bleeding esophageal varices and HRS type 1 and is usually administered using multiple IV doses given by bolus injections in the hospital.

This study is an open label, first in human study of PHIN-214. PHIN-214 is a terlipressin derivative administered subcutaneously. It is a partial V1a agonist which is designed to reduce splanchnic blood pooling and portal hypertension. A resultant increase in systemic pressure and renal arterial pressure may increase kidney perfusion and creatinine clearance.

This study will evaluate a single dose of PHIN-214 (in Part 1) and in Part 2, daily doses of PHIN-214 for up to 28-days (called multiple ascending doses) of PHIN-214 to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of PHIN-214 in subjects with advanced cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

1. History of cirrhosis based on histology or a combination of clinical, radiological, or biochemical assessment and classified as Child-Pugh A or B
2. Participants may be male or female aged 18 to 75 years.
3. Body mass index (BMI) within the range 18 to 40 kg/m2 (inclusive) at screening.
4. Female participants must be non-pregnant, non-lactating, or of non-childbearing potential or using highly efficient contraception for the full duration of the study

Key Exclusion Criteria:

1. Significant abnormalities in medical history or on physical examination, including: respiratory disease requiring therapy or history of respiratory failure, cardiovascular disease or hypertension, electrocardiogram abnormalities or history of significant EKG abnormalities.
2. History of diabetes insipidus, syndrome of inappropriate antidiuretic hormone secretion, or any other disorder associated with fluid or sodium imbalance.
3. Significant kidney disease
4. Hepatic encephalopathy (HE) or altered mental status requiring hospitalization; variceal bleeding or upper gastrointestinal bleeding; or type 1 hepatorenal syndrome with acute kidney injury (HRS-AKI) during the previous 3 months prior to Screening.
5. Acute-on-chronic liver failure.
6. Recipient of a patent transjugular intrahepatic portosystemic shunt (TIPS).
7. Known positive HIV serology confirmed by HIV viral load.
8. Subjects with acute infections, including acute viral hepatitis (subjects with chronic hepatitis B are eligible if treatment regimen is stable ≥ 3 months prior to study inclusion).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose or optimal beneficial dose of PHIN-214 in multiple ascending dose; safety and tolerability. | may be up to six weeks
  Incidence of adverse effects (type and severity), incidence of dose limiting toxicities, changes in key laboratory measures
Pharmacokinetics of PHIN-214 | up to six weeks
  plasma concentration of PHIN-214
Pharmacokinetics of PHIN-214 metabolite | up to six weeks
  plasma concentration of PHIN-214 metabolite

SECONDARY OUTCOMES:
Immunogenicity of PHIN-214 | up to six weeks
  anti-drug antibody testing

OTHER OUTCOMES:
Blood pressure | up to six weeks
  Blood pressure (vital signs)
Heart rate | up to six weeks
  Heart rate (vital signs)
12-lead ECG | up to six weeks
  12-lead ECG
Oxygenation level | up to six weeks
  Oxygenation level by pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia C Jones, Study Chair — PharmaIN
Locations (9):
- United States (9):
  - Arizona Liver Health, Chandler, Arizona
  - Southern California Research Center, Coronado, California
  - Tandem Clinical Research, Marrero, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Methodist Health System, Dallas Medical Center, Dallas, Texas
  - VA North Texas Healthcare System, Dallas, Texas
  - Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided